CLINICAL TRIAL: NCT00172198
Title: A Prospective, Controlled, Randomized, Study Evaluating the Clinical Efficacy, Including Nutritional Status, Immune Function and Safety of Omegaven (w-3 Fish Oil) Supplemented Parenteral Nutrition in Subjects of SICU.
Brief Title: Omegaven (w-3 Fish Oil) Supplemented Parenteral Nutrition in Subjects of SICU.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 183CL1
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2005-09-15 (Estimated); Status verified 2005-01

CONDITIONS: Critical Ill Patients in SICU
Keywords: w-3 fish oil; Nutrition; immune; intensive care; patients

INTERVENTIONS:
Drug: Omegaven 10%

SUMMARY:
1. A prospective, controlled, randomized, study evaluating the clinical efficacy, including nutritional status, immune function and safety of Omegaven (ω-3 fish oil) supplemented parenteral nutrition in subjects of SICU.
2. Study patients are the critical ill patients in SICU of NTUH and the enrolled patients will be 30 subjects ,including 15 in each treatment group.
3. During parenteral nutrition, fat emulsions will be given separately from amino acid and glucose solutions. Infusion pump must be used.The recommended infusion duration of the daily lipid emulsion is 16 hours (0.0625 g fat/kg B.W./hour) from 8:00 am to 12:00 pm.
4. During the study the assessments of safety and efficacy are to be performed according to case report form. The assessment for safety variables including blood pressure、heat rate 、body temperature、liver function、renal function、coagulation、WBC、lipid profile etc. In addition，the assessments for efficacy variables including lymphocytes、cytokines(IL-1、IL-2、IL-6、IL-8、IL-11、IL-18、OX40 ligand、G-CSF、FN-γ、TGF-β1、TNF-α etc)、incidence of infections、 length of ICU and hospital stay、mortality etc.

DETAILED DESCRIPTION:
1. A prospective, controlled, randomized, study evaluating the clinical efficacy, including nutritional status, immune function and safety of Omegaven (ω-3 fish oil) supplemented parenteral nutrition in subjects of SICU.
2. Study patients are the critical ill patients in SICU of NTUH and the enrolled patients will be 30 subjects ,including 15 in each treatment group.
3. During parenteral nutrition, fat emulsions will be given separately from amino acid and glucose solutions. Infusion pump must be used.The recommended infusion duration of the daily lipid emulsion is 16 hours (0.0625 g fat/kg B.W./hour) from 8:00 am to 12:00 pm.
4. During the study the assessments of safety and efficacy are to be performed according to case report form. The assessment for safety variables including blood pressure、heat rate 、body temperature、liver function、renal function、coagulation、WBC、lipid profile etc. In addition，the assessments for efficacy variables including lymphocytes、cytokines(IL-1、IL-2、IL-6、IL-8、IL-11、IL-18、OX40 ligand、G-CSF、FN-γ、TGF-β1、TNF-α etc)、incidence of infections、 length of ICU and hospital stay、mortality etc.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients between 15 and 75 years of age
* Expected ICU stay and TPN support requirement > 7 days
* Hemodynamically stable
* Serum bilirubin < 2.5 mg/dl
* Serum creatinine < 1.4 mg/dl
* INR (international Normalized ratio of PT) < 1.4
* Written informed consent from the subject

Exclusion Criteria:

* Pregnant or lactating women. (Pre-menopause women, capable of bearing children will undergo pregnancy test)
* General contraindications of infusion therapy; acute pulmonary oedema,hyperhydration and decompensated cardiac insufficiency
* Known hypersensitivity to egg- or soy protein or any of the ingredients
* Severe blood coagulation disorders
* Shock necessitating acute resuscitation at the discretion of the investigator
* Diabetes mellitus with known ketoacidosis within 7 days of onset of study treatment
* APACHE II score > 25
* Renal insufficiency defined as serum creatinine value of >1.4 mg/dl
* Subjects with severe liver dysfunction which contraindicates the use of parenteral nutrition at the discretion of the investigator
* Known type IV hyperlipidemia, disturbances in lipid metabolism or hypertriglyceridemia (at the time of inclusion, a blood sample (fasting) for serum triglyceride assessment has to be taken. The sample has to be analysed before start of trial treatment. In case of fasting serum triglyceride value of >4 mmol/l (>354 mg/dl) the subject must be withdrawn.
* Unconscious or uncooperative patients
* Participation in a clinical study with an investigational drug or an investigational medical device within one month prior to start of study

Ages: 15 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30
Dates: Start 2005-03; Study Completion 2007-03

PRIMARY OUTCOMES:
Lymphocytes:T4,T8,B,T,NK
Cytokine secretion:IL-1、IL-2、IL-6、IL-8、IL-11、IL-18、OX40 ligand、G-CSF、FN-γ、TGF-β1、TNF-α.
Clinical outcome:incidence of infections,length of ICU and hospital stay,ventilation,mortality

SECONDARY OUTCOMES:
Liver function(AST,ALT,bilirubin,ALP,rGT,albumin)
renal function(BUN,creatinine)
AC blood sugar
coagulation(INR,aPTT)
sodium
potassium
chloride
calcium
magnesium
phosphate
total white blood cell counts
platelets
haemoglobin
haematoc

CONTACTS AND LOCATIONS:
Overall Officials: Hong-Shiee Lai, Professor, Principal Investigator — National Taiwan University Hospital, Taipei, Taiwan
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Background] Roulet M, Frascarolo P, Pilet M, Chapuis G. Effects of intravenously infused fish oil on platelet fatty acid phospholipid composition and on platelet function in postoperative trauma. JPEN J Parenter Enteral Nutr. 1997 Sep-Oct;21(5):296-301. doi: 10.1177/0148607197021005296. PMID 9323693